CLINICAL TRIAL: NCT01203631
Title: A Randomised, Double-blind, Parallel-group, Placebo Controlled Induction Trial to Assess the Clinical Efficacy and Safety of NNC 0142-0000-0002 in Subjects With Moderately to Severely Active Crohn's Disease
Brief Title: Safety and Efficacy of NNC 0142-0000-0002 in Subjects With Moderately to Severely Active Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8555-3797; 2010-020836-21 (EudraCT Number); U1111-1116-2695 (Other: WHO)
Record Dates: First submitted 2010-09-15; First posted 2010-09-16 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Inflammation; Crohn's Disease
MeSH Terms: conditions — Inflammation; Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC 0142-0000-0002 (Experimental)
  Interventions: Drug: NNC 0142-0000-0002
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NNC 0142-0000-0002 — A single dose administered subcutaneously (s.c., under the skin)
  Arms: NNC 0142-0000-0002
Drug: Placebo — A single dose administered subcutaneously (s.c., under the skin)
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe and North America. The aim of the trial is to assess disease activity and safety in subjects with moderately to severely active Crohn's disease (CD) when treated with NNC 0142-0000-0002.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with CD for at least 3 months
* Subjects not treated before, or subjects who have either not responded to treatment, or responded and then lost the response during continued administration of a therapeutic compound

Exclusion Criteria:

* Any of the following: Symptomatic bowel obstruction, short bowel syndrome, ileostomy or colostomy, surgical bowel resection within 6 months prior to randomisation or clinically relevant un-drained abscess
* History of dysplasia or malignancy in the colon
* Any ongoing chronic or active infectious disease or microbial infection requiring systemic oral or intravenous treatment against infection within 1 month prior to randomisation
* Body mass index (BMI) higher or equal to 38.0 kg/m^2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Change in disease activity assessed by CDAI (Crohn's disease activity index) | From baseline to week 4

SECONDARY OUTCOMES:
Number of adverse events (AEs) | From baseline to weeks 12 and 24
Immunogenicity of NNC 142-0002 | At week 24

CONTACTS AND LOCATIONS:
Overall Officials: Najat EL Bariaki, Study Director — Novo Nordisk A/S
Locations (23):
- United States (16):
  - Novo Nordisk Clinical Trial Call Center, Anaheim, California
  - Novo Nordisk Clinical Trial Call Center, Lakewood, Colorado
  - Novo Nordisk Clinical Trial Call Center, Chicago, Illinois
  - Novo Nordisk Clinical Trial Call Center, Louisville, Kentucky
  - Novo Nordisk Clinical Trial Call Center, Annapolis, Maryland
  - Novo Nordisk Clinical Trial Call Center, Chevy Chase, Maryland
  - Novo Nordisk Clinical Trial Call Center, Towson, Maryland
  - Novo Nordisk Clinical Trial Call Center, Chesterfield, Michigan
  - Novo Nordisk Clinical Trial Call Center, Troy, Michigan
  - Novo Nordisk Clinical Trial Call Center, New York, New York
  - Novo Nordisk Clinical Trial Call Center, Asheville, North Carolina
  - Novo Nordisk Clinical Trial Call Center, Fayetteville, North Carolina
  - Novo Nordisk Clinical Trial Call Center, Raleigh, North Carolina
  - Novo Nordisk Clinical Trial Call Center, Germantown, Tennessee
  - Novo Nordisk Clinical Trial Call Center, Charlottesville, Virginia
  - Novo Nordisk Clinical Trial Call Center, Milwaukee, Wisconsin
- Leuven, Belgium
- Edmonton, Alberta, Canada
- Paris, France
- Győr, Hungary
- Kfar Saba, Israel
- Warsaw, Poland
- Saint Petersburg, Russia

REFERENCES:
- [Derived] Allez M, Skolnick BE, Wisniewska-Jarosinska M, Petryka R, Overgaard RV. Anti-NKG2D monoclonal antibody (NNC0142-0002) in active Crohn's disease: a randomised controlled trial. Gut. 2017 Nov;66(11):1918-1925. doi: 10.1136/gutjnl-2016-311824. Epub 2016 Aug 3. PMID 27489241
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com